CLINICAL TRIAL: NCT04270864
Title: A Phase I Trial Assessing the Safety and Efficacy of an Anti-tumor Immunity Priming Strategy Combining Intratumoral Tilsotolimod, a TLR-9 Agonist, Together With Intratumoral Ipilimumab and Intravenous Nivolumab in Patients With Advanced Cancers
Brief Title: Intratumoral Tilsotolimod, a TLR-9 Agonist, Together With Intratumoral Ipilimumab and Intravenous Nivolumab in Patients With Advanced Cancers
Acronym: PRIMO
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The part A of the trial has been completed according to the protocol. The part B has not been opened because of unfeasibility (experimental products not yet available).
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-004790-26; 2019/2840 (Other: CSET number)
Record Dates: First submitted 2020-02-10; First posted 2020-02-17 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Advanced Cancer
MeSH Terms: interventions — Ipilimumab; Nivolumab; tilsotolimod

STUDY DESIGN:
Intervention Model Description: Open label, phase Ib study of intratumoral tilsotolimod in combination with intratumoral ipilimumab and intravenous nivolumab.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Regimen A1 (Experimental): Combination between nivolumab IV Q3W and dual intratumoral injections of Ipilimumab and Tilsotolimod Q3W
  Interventions: Drug: Ipilimumab; Drug: Nivolumab; Drug: Tilsotolimod
- Regimen A2 (Experimental): Combination between nivolumab IV Q3W and dual intratumoral injections of Ipilimumab and Tilsotolimod QW
  Interventions: Drug: Ipilimumab; Drug: Nivolumab; Drug: Tilsotolimod

INTERVENTIONS:
Drug: Ipilimumab — 20mg (4mL) IT
Drug: Nivolumab — 360mg IV then 480mg IV
Drug: Tilsotolimod — 8 mg (2mL) IT

SUMMARY:
Open label, phase Ib study of intratumoral tilsotolimod in combination with intratumoral ipilimumab and intravenous nivolumab.

The trial will be divided into two parts:

PART A:

the first part will assess the safety of two regimen and will recruit patients with all types of injectable solid malignancies

PART B:

the second part will include 3 expansion cohorts of 15 patients:

* B1: anti-PD-1 refractory advanced NSCLC cohort
* B2: anti-PD-1 refractory advanced melanoma cohort
* B3: immunotherapy naïve microsatellite stable colorectal cancer (MSS CRC) cohort

ELIGIBILITY:
Inclusion Criteria:

1. Men and women ≥ 18 years of age
2. Patient should understand, sign, and date the written informed consent form prior to any protocol-specific procedures performed.
3. For part A & B: patients must have a histologically confirmed and clinically or radiologically progressing unresectable advanced cancers relapsing or refractory after conventional therapies. Patients pre-treated with immunotherapy are eligible if they have not developed treatment-related CTCAE v.5 grade ≥ 4 irAE or any grade ≥ 3 irAE lasting for more than 21 days. However, patients who developed auto-immune endocrinopathies during previous immunotherapy and are well treated with hormone substitutive therapy do not fell into this category and should remain eligible.
4. For part B (expansion cohorts):

   1. For part B1: histologically confirmed and clinically or radiologically progressing unresectable Stage III or Stage IV NSCLC, with a history of pre-treatment by anti-PD-1. Patients should have a clinically or radiologically documented disease progression after having either:

      1. received an anti-PD-1 monotherapy first line followed by a chemotherapy second line
      2. or a combination of anti-PD-1 + chemotherapy first line
   2. For B2 cohort: histologically confirmed and clinically or radiologically progressing unresectable Stage III or Stage IV melanoma, as per AJCC staging system, naïve of anti-PD-(L)1 and/or anti-CTLA-4 (ocular melanoma excluded).
   3. For part B3: histologically confirmed and clinically or radiologically progressing unresectable Stage III or Stage IV MSS CRC cancer naïve of anti-PD(L)1 and anti-CTLA4 therapy . Patients must have received or must be ineligible to standard treatments (chemotherapy with 5-FU, oxaliplatin, irinotecan ; bevacizumab ; anti-EGFR therapies if applicable).
5. Patient with at least one injectable tumor lesion (largest diameter ≥1cm; smallest diameter ≥1,5cm if lymph node) which is measurable as per RECIST 1.1 criteria and which will be used as the intratumoral immunotherapy priming site. Patients with additional tumor lesions should be monitored for both injected and non-injected lesions as per iRECIST criteria. Patients with additional peritoneal carcinomatosis or pleural tumoral effusions or other tumoral involvement could be included if they can be evaluable by an objective criteria such as PET-scan or tumor marker or ctDNA.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
7. Treatment naïve subjects or patients relapsing after prior local or systemic anticancer therapy. Note that systemic anticancer therapy is permitted if it was completed at least 28 days or 5 times its half-life (whichever is shorter) prior to the first study dose, and all clinically significant related adverse events have either returned to baseline or stabilized. Treatment naïve patients are allowed if they are unsuitable for conventional therapy.
8. Measurable disease by CT or MRI per RECIST 1.1 criteria.
9. Patients willing to undergo intratumoral injections and tumor biopsies. Biopsies and intratumoral injections should be performed without any pain. Local anesthesia should be performed if necessary prior any intratumoral injection/biopsy. If a patient needs to undergo a systemic sedation or anesthesia for his intratumoral biopsies/injections, this should be validated during the screening phase by a consultation with an anesthesist from the team who would be in charge of such procedure.
10. Prior radiotherapy must have been completed at least 2 weeks prior to study drug administration. Irradiated lesion should not be chosen as injectable nor target lesion.
11. Screening laboratory values must meet the following criteria and should be obtained within 14 days prior to randomization:

    * Neutrophils to Lymphocytes Ratio (NLR) ≤ 6*
    * Platelets ≥ 100 x103/μL
    * Hemoglobin ≥ 8.0 g/dL (transfusion allowed)
    * Serum creatinine ≤ 1.5 x ULN or creatinine clearance (CrCl) > 40mL/min (using the Cockcroft-Gault formula)
    * ALT ≤3.0 x upper limit of normal (ULN); if liver metastases ALT ≤5.0 x ULN
    * Total Bilirubin <1.5 x ULN (except subjects with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL).
    * LDH ≤ Upper Limit of Normal (ULN)
    * Albumin ≥ Lower Limit of Normal (LLN)
12. Subject Re-enrollment: This study permits the re-enrollment of a subject that has discontinued the study as a screening failure (ie, subject has not been treated) after obtaining agreement from the medical coordinator prior to re-enrolling a subject. If reenrolled, the subject must be re-consented.
13. Women of childbearing potential (WOCBP) must have a negative urine or serum β-HCG pregnancy test within 24 hours prior to initiation of treatment. Sexually active female patients must agree to use two methods of effective contraception, one of them being a barrier method, or to abstain from sexual activity during the study and for at least 5 months after last study drug administration. Sexually active males patients (and their female partners) must agree to use two methods of effective contraception, one of them being a barrier method, or to abstain from sexual activity during the study and for at least 7 months after last study drug administration.
14. Patients must be willing and able to comply with the visits, treatments, procedures, and laboratory tests, and other requirements that are scheduled in the protocol.
15. Patients must be affiliated to a social security system or beneficiary of the same

Exclusion Criteria:

1. Active brain metastases or leptomeningeal metastases. Subjects with brain metastases or leptomeningeal disease are eligible if these lesions have been treated or if they are asymptomatic without any steroids and there is no clinical evidence of progression within 14 days prior to first dose of study drug administration. CNS lesions should be monitored by contrast enhanced MRI at disease assessment timepoints.
2. Any serious or uncontrolled medical disorder that, in the opinion of the investigator, may increase the risk associated with study participation or study drug administration, impair the ability of the subject to receive protocol therapy, or interfere with the interpretation of study results.
3. Prior malignancy active within the previous 3 years except for Lynch syndrome patients and locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast.
4. Subjects with active, known or suspected autoimmune disease including a history of anti-phospholipid syndrome. Subjects with vitiligo, type I diabetes mellitus, auto-immune endocrinopathy only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
5. Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids, and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
6. Part B: Prior treatment with an anti-PD-1, anti-PD-L1, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell costimulation or immune checkpoint pathways, except for the NSCLC expansion cohort.
7. Positive test for human immunodeficiency virus (HIV) or known acquire immunodeficiency syndrome (AIDS) unless the viral load is well controlled by anti-retroviral therapy and the CD4+ T-cell count remained beyond 500/mm3 for the last 6 months.
8. Positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV antibody) indicating acute or chronic infection.
9. History of allergy to study drug components.
10. History of severe hypersensitivity reaction to any monoclonal antibody.
11. Pregnancy or breastfeeding
12. Patients presenting coagulation abnormalities and/or patients requiring concomitant treatment with therapeutic doses of anticoagulants. Prophylactic low dose of anticoagulants for thrombo-embolic events is allowed. Prophylactic anticoagulants shall be stopped during 24h prior and after deep lesion biopsies/injections. No stopping rule for biopsies/injections of skin and sub-cutaneous lesions. Up to 150mg/d aspirin monotherapy allowed.
13. No live vaccines while on study treatment and for at least 6 months afterwards. Live vaccines include rubella, mumps, measles, BCG, yellow fever and shingles vaccine.For other types of vaccines, a minimum of 28 days between the last vaccine and study treatment is required.
14. During participation in this study, patients will not receive any other clinical investigational drugs or any other anti-tumor drugs.
15. Patient under guardianship or deprived of his liberty by a judicial or administrative decision or incapable of giving its consent.
16. Tumor lesions presenting with intracavitary overflow in the pleural or peritoneal space are not eligible for intratumoral injections.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-04-10 (Actual); Primary Completion 2021-07-13 (Actual); Study Completion 2023-09-25 (Actual)

PRIMARY OUTCOMES:
Describe the incidence of Dose-intensity limiting toxicities | during a 28 days period after Cycle 1Day 1 (each cycle is 28 days)

CONTACTS AND LOCATIONS:
Locations (1):
- Gustave Roussy, Villejuif, Val De Marne, France

IPD SHARING:
Plan to Share IPD: Yes